CLINICAL TRIAL: NCT02862574
Title: Evaluation of the Efficacy and Safety of GS-5745 as Add-On Therapy to a Tumor Necrosis Factor Inhibitor and Methotrexate Regimen in Subjects With Moderate to Severe Rheumatoid Arthritis
Brief Title: Andecaliximab as Add-On Therapy to a Tumor Necrosis Factor Inhibitor and Methotrexate Regimen in Adults With Moderately to Severely Active Rheumatoid Arthritis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated by sponsor and decision was not due to any safety signals.
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-373-1499; 2016-000897-39 (EudraCT Number)
Record Dates: First submitted 2016-08-08; First posted 2016-08-11 (Estimated); Results first posted 2018-06-27 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-05

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Tumor Necrosis Factor Inhibitor; TNF-IR; Methotrexate
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — andecaliximab; Methotrexate; Tumor Necrosis Factor Inhibitors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Andecaliximab 300 mg (Experimental): Andecaliximab 300 mg for 12 weeks, in addition to their current regimen of a TNF inhibitor and methotrexate.
  Interventions: Drug: Andecaliximab; Drug: Methotrexate; Drug: TNF Inhibitor
- Andecaliximab 150 mg (Experimental): Andecaliximab 150 mg + placebo for 12 weeks, in addition to their current regimen of a TNF inhibitor and methotrexate.
  Interventions: Drug: Andecaliximab; Drug: Placebo; Drug: Methotrexate; Drug: TNF Inhibitor
- Placebo (Placebo Comparator): Placebo weekly for 12 weeks, in addition to their current regimen of a TNF inhibitor and methotrexate.
  Interventions: Drug: Placebo; Drug: Methotrexate; Drug: TNF Inhibitor
- Open-Label Extension (Experimental): On the Week 12 visit, eligible participants may choose to participate in the open-label portion of the study to receive open-label andecaliximab 300 mg for 52 weeks, in addition to their current regimen of a TNF inhibitor and methotrexate.
  Interventions: Drug: Andecaliximab; Drug: Methotrexate; Drug: TNF Inhibitor

INTERVENTIONS:
Drug: Andecaliximab — Administered via subcutaneous injection once weekly
  Other Names: GS-5745
  Arms: Andecaliximab 150 mg; Andecaliximab 300 mg; Open-Label Extension
Drug: Placebo — Administered via subcutaneous injection once weekly
  Arms: Andecaliximab 150 mg; Placebo
Drug: Methotrexate — Administered orally weekly as part of the participant's current treatment regimen
Drug: TNF Inhibitor — An approved stable subcutaneous formulation of one of the following TNF inhibitors may include adalimumab, certolizumab, etanercept, or golimumab.

SUMMARY:
The primary objective of this study is to evaluate the efficacy of andecaliximab (GS-5745) versus placebo as an add-on therapy to a tumor necrosis factor (TNF) inhibitor and methotrexate in adults with moderate to severe rheumatoid arthritis (RA).

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of RA (according to the 2010 American College of Rheumatology and European League Against Rheumatism (ACR/EULAR) classification criteria) confirmed at screening
* Must have taken oral or parenteral methotrexate (MTX) dosed from 7.5 to 25 mg/week continuously for at least 12 weeks and tolerated this medication, with at least 6 weeks of stable dose (defined as no change in prescription) prior to first dose of study drug
* Individuals on MTX may also be on concurrent chloroquine or hydroxychloroquine at a stable dose (defined as no change in prescription) for at least 4 week prior to Baseline; if so, they should plan to continue this medication for the duration of the study
* Must have an inadequate response to ≥ 12 weeks of ongoing treatment with an approved, stable subcutaneous (SC) formulation of TNF inhibitor (adalimumab, certolizumab pegol, etanercept, or golimumab), or marketed SC biosimilar TNF inhibitor with at least 6 weeks of stable dose (defined as no change in prescription), defined as: must have a DAS28(CRP) > 3.2 at screening AND must have ≥ 3 swollen and ≥ 3 tender joints (using the DAS28 joint counts) at screening and at baseline (do not need to be the same joints)
* Non-steroidal anti-inflammatory drugs (NSAIDs) and/or oral corticosteroids (≤ 10 mg prednisone/day or equivalent) at a stable dose (defined as no change in prescription) for ≥ 4 weeks prior to baseline are allowed and throughout the blinded period of the study. PRN NSAID for indications other than RA are also allowed. (PRN means "pro re nata" or when necessary)
* Tuberculosis (TB) Screening: Must meet either a. or b.:

  1. A negative history of TB infection and a negative QuantiFERON® TB-Gold In-Tube test and chest x-ray results. (QuantiFERON® tests with inconclusive results may be repeated one time. If the repeat result is also inconclusive, the individual will be excluded from the study).

     OR,
  2. Individuals with a history of latent TB treated with a full course of prophylaxis as per local guidelines are allowed per investigator judgment. It is the responsibility of the investigator to verify the adequacy of previous treatment and to provide appropriate documentation. In these cases, no QuantiFERON® test need be obtained. In addition, these cases must be approved by the medical monitor prior to enrollment. (Any new diagnosis of latent TB or prior untreated /partially treated latent TB in NOT allowed (ie, individuals who require prophylactic therapy for TB during the study). Any prior history of active TB [regardless of treatment] is exclusionary).
* A negative chest x-ray (views per local guidelines) for active TB or other lung disease at screening; or a chest x-ray within 90 days of screening if films or report are available for investigator review

Key Exclusion Criteria:

* Current treatment with any other disease modifying anti-rheumatic drug (DMARD) other than MTX, chloroquine or hydroxychloroquine, OR current treatment with other immune modulating/suppressive non-biologic and biologic medications as described in the study protocol
* Intraarticular corticosteroid injection of any joint within 4 weeks of baseline
* Any infection requiring oral antimicrobial therapy within 2 weeks prior to baseline
* Current inflammatory joint disease, other than RA, such as gout, reactive arthritis, psoriatic arthritis, seronegative spondylarthritis, or Lyme disease, OR other current autoimmune diseases such as: systemic lupus erythematosus (SLE), inflammatory bowel disease, fibromyalgia, polymyalgia rheumatica, scleroderma, inflammatory myopathy, mixed connective tissue disease, or other overlap syndrome that would interfere with the evaluation of RA or require protocol prohibited medication (individuals with Sjogren's syndrome or controlled thyroiditis as defined by the investigator are not excluded)
* Active systemic involvement secondary to RA such as vasculitis or Felty's syndrome
* History of any of the following within 12 months of baseline:

  * infection requiring parenteral antibiotics or hospitalization
  * any life-threatening infection
  * sepsis
* The results of the following laboratory tests performed at the central laboratory at screening meet any of the criteria below:

  * Hemoglobin < 8.0 g/dL (International System of Units (SI): < 80 g/L)
  * White blood cells < 3.0 x 10^3 cells/mm^3 (SI: < 3.0 x 10^9 cells/L)
  * Neutrophils < 1.5 x 10^3 cells/mm^3 (SI: < 1.5 x 10^9 cells/L)
  * Lymphocytes < 0.5 x 10^3 cells/mm^3 (SI: < 0.5 x 10^9 cells/L)
  * Platelets < 100 x 10^3 cells/mm^3 (SI: < 100 x 10^9 cells/L)
  * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 2 x upper limit of normal (ULN)
  * Total bilirubin level ≥ 2 x ULN unless the individual has been diagnosed with Gilbert's disease and this is clearly documented
  * Estimated glomerular filtration rate < 40 mL/min/1.73 m^2 based on the Modification of Diet in Renal Disease (MDRD) formula
  * Positive HIV serology during screening
  * Evidence of active Hepatitis B Virus (HBV) infection
  * Evidence of active Hepatitis C Virus (HCV) infection
* Any uncontrolled clinically significant laboratory abnormality that would affect interpretation of study data or the individual's participation in the study
* Malignancy or a history of malignancy or lymphoproliferative disorder within 10 years of screening with the following exceptions:

  * Carcinoma in situ of the cervix that has been successfully treated
  * Adequately treated basal or squamous cell cancer that has been successfully treated

Note: Other protocol defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2017-06-26 (Actual); Study Completion 2017-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (8):
- United States (8):
  - Stanford University, Palo Alto, California
  - Omega Research Consultants, LLC, DeBary, Florida
  - G. Timothy Kelly, MD, Las Vegas, Nevada
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Albuquerque Center for Rheumatology, Albuquerque, New Mexico
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Tekton Research, Austin, Texas
  - Accurate Clinical Research, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States. The first participant was screened on 15 December 2016. The last study visit occurred on 07 August 2017.
Pre-assignment Details: 28 participants were screened.
Groups:
- Andecaliximab 300 mg: Double-Blind Period: Andecaliximab 300 mg administered via subcutaneous injection once weekly for 12 weeks, in addition to participant's current regimen of a tumor necrosis factor (TNF) inhibitor and methotrexate
  Open-Label Period: Andecaliximab 300 mg administered via subcutaneous injection once weekly for up to 52 weeks, in addition to participant's current regimen of a TNF inhibitor and methotrexate
- Andecaliximab 150 mg: Double-Blind Period: Andecaliximab 150 mg administered via subcutaneous injection + placebo once weekly for 12 weeks, in addition to participant's current regimen of a TNF inhibitor and methotrexate
  Open-Label Period: Andecaliximab 300 mg administered via subcutaneous injection once weekly for up to 52 weeks, in addition to participant's current regimen of a TNF inhibitor and methotrexate
- Placebo: Double-Blind Period: Placebo administered via subcutaneous injection once weekly for 12 weeks, in addition to participant's current regimen of a TNF inhibitor and methotrexate
  Open-Label Period: Andecaliximab 300 mg administered via subcutaneous injection once weekly for up to 52 weeks, in addition to participant's current regimen of a TNF inhibitor and methotrexate
Period: Double-Blind Treatment Period
Arm/Group | Andecaliximab 300 mg | Andecaliximab 150 mg | Placebo
Started | 5 | 5 | 5
Completed | 2 | 3 | 1
Not Completed | 3 | 2 | 4
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Study Terminated by Sponsor | 3 | 1 | 4
Period: Open-Label Treatment Period
Arm/Group | Andecaliximab 300 mg | Andecaliximab 150 mg | Placebo
Started | 2 | 3 | 1
Completed | 0 | 0 | 0
Not Completed | 2 | 3 | 1
Not completed — Study Terminated by Sponsor | 2 | 3 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who received at least 1 dose of study drug
Groups:
- Andecaliximab 300 mg: Double-Blind Period: Andecaliximab 300 mg administered via subcutaneous injection once weekly for 12 weeks, in addition to participant's current regimen of a TNF inhibitor and methotrexate
  Open-Label Period: Andecaliximab 300 mg administered via subcutaneous injection once weekly for up to 52 weeks, in addition to participant's current regimen of a TNF inhibitor and methotrexate
- Total: Total of all reporting groups
Arm/Group | Andecaliximab 300 mg | Andecaliximab 150 mg | Placebo | Total
Number analyzed (Participants) | 5 | 5 | 5 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (16.3) | 57 (9.3) | 58 (5.6) | 56 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 4 | 11
  Male | 2 | 1 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 2
  Not Hispanic or Latino | 5 | 3 | 5 | 13
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 1 | 3
  White | 3 | 5 | 4 | 12
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Disease Activity Score C-reactive Protein (DAS28(CRP)) [Mean (Standard Deviation); unit: units on a scale] — The DAS28 score is a measure of the participant's disease activity calculated using the tender joint counts (28 joints), swollen joint counts (28 joints), Patient's Global Assessment of Disease Activity (visual analog scale: 0 = no disease activity to 100 = maximum disease activity), and C-Reactive Protein (CRP) for a total possible score of 2 to 10. Higher values indicate higher disease activity.
  units on a scale | 5.79 (0.814) | 5.90 (0.752) | 5.69 (0.887) | 5.79 (0.764)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in DAS28(CRP) at Week 12
Description: The DAS28 score is a measure of the participant's disease activity calculated using the tender joint counts (28 joints), swollen joint counts (28 joints), Patient's Global Assessment of Disease Activity (visual analog scale: 0 = no disease activity to 100 = maximum disease activity), and CRP for a total possible score of 1 to 9.4. Higher values indicate higher disease activity. A negative change from baseline indicates improvement.
Time Frame: Baseline; Week 12
Population: Participants in the Full Analysis Set (all randomized participants who received at least 1 dose of study drug) with available data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Andecaliximab 300 mg: Andecaliximab 300 mg administered via subcutaneous injection once weekly for 12 weeks, in addition to participant's current regimen of a TNF inhibitor and methotrexate
- Andecaliximab 150 mg: Andecaliximab 150 mg administered via subcutaneous injection + placebo once weekly for 12 weeks, in addition to participant's current regimen of a TNF inhibitor and methotrexate
- Placebo: Placebo administered via subcutaneous injection once weekly for 12 weeks, in addition to participant's current regimen of a TNF inhibitor and methotrexate
Arm/Group | Andecaliximab 300 mg | Andecaliximab 150 mg | Placebo
Number analyzed (Participants) | 2 | 3 | 3
units on a scale | 0.13 (0.115) | -1.51 (0.670) | -0.36 (0.353)

2. Secondary Outcome: Percentage of Participants That Achieve DAS28(CRP) ≤ 3.2 at Week 12
Description: as for outcome 1
Time Frame: Week 12
Population: Full Analysis Set: all randomized participants who received at least 1 dose of study drug
Measure: Number; unit: percentage of participants
Arm/Group | Andecaliximab 300 mg | Andecaliximab 150 mg | Placebo
Number analyzed (Participants) | 5 | 5 | 5
percentage of participants | 0 | 0 | 0

3. Secondary Outcome: Percentage of Participants That Achieve DAS28(CRP) < 2.6 at Week 12
Description: as for outcome 1
Time Frame: Week 12
Population: Full Analysis Set: all randomized participants who received at least 1 dose of study drug
Measure: Number; unit: percentage of participants
Arm/Group | Andecaliximab 300 mg | Andecaliximab 150 mg | Placebo
Number analyzed (Participants) | 5 | 5 | 5
percentage of participants | 0 | 0 | 0

4. Secondary Outcome: Plasma Concentration of Andecaliximab
Description: The plasma concentrations of andecaliximab were not collected and were not analyzed.
Time Frame: Day 4 or 6 (± 1 day)
Arm/Group | Andecaliximab 300 mg | Andecaliximab 150 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to the last dose date (maximum: 127 days) plus 30 days
Description: Safety Analysis Set: participants who received at least 1 dose of study drug
Groups:
- Andecaliximab 300 mg (Double-Blind): Andecaliximab 300 mg administered via subcutaneous injection once weekly for 12 weeks, in addition to participant's current regimen of a TNF inhibitor and methotrexate
- Andecaliximab 150 mg (Double-Blind): Andecaliximab 150 mg administered via subcutaneous injection + placebo once weekly for 12 weeks, in addition to participant's current regimen of a TNF inhibitor and methotrexate
- Placebo (Double-Blind): Placebo administered via subcutaneous injection once weekly for 12 weeks, in addition to participant's current regimen of a TNF inhibitor and methotrexate
- Andecaliximab 300 mg (Open-Label): Andecaliximab 300 mg administered via subcutaneous injection once weekly for up to 52 weeks, in addition to participant's current regimen of a TNF inhibitor and methotrexate
Arm/Group | Andecaliximab 300 mg (Double-Blind) | Andecaliximab 150 mg (Double-Blind) | Placebo (Double-Blind) | Andecaliximab 300 mg (Open-Label)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 1/6
Other Adverse Events (participants affected / at risk) | 3/5 | 2/5 | 2/5 | 2/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Andecaliximab 300 mg (Double-Blind) (N=5) | Andecaliximab 150 mg (Double-Blind) (N=5) | Placebo (Double-Blind) (N=5) | Andecaliximab 300 mg (Open-Label) (N=6)
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Andecaliximab 300 mg (Double-Blind) (N=5) | Andecaliximab 150 mg (Double-Blind) (N=5) | Placebo (Double-Blind) (N=5) | Andecaliximab 300 mg (Open-Label) (N=6)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Gilead decided to discontinue the development of andecaliximab in RA and this study was terminated. The decision was not due to any safety concerns. Because only 15 participants were enrolled, no formal statistical testing was completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (4):
  • Study Protocol: Original (2016-03-14): https://cdn.clinicaltrials.gov/large-docs/74/NCT02862574/Prot_000.pdf
  • Study Protocol: Amendment 1 (2016-06-24): https://cdn.clinicaltrials.gov/large-docs/74/NCT02862574/Prot_001.pdf
  • Study Protocol: Amendment 2 (2016-09-23): https://cdn.clinicaltrials.gov/large-docs/74/NCT02862574/Prot_002.pdf
  • Statistical Analysis Plan (2017-12-11): https://cdn.clinicaltrials.gov/large-docs/74/NCT02862574/SAP_003.pdf